CLINICAL TRIAL: NCT04906213
Title: CardioRenal Effects of SGLT2 Inhibition in Kidney Transplant Recipients
Acronym: CREST-KT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study closed per PI decision due to poor accrual since 2022.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Pro00107752
Record Dates: First submitted 2021-05-18; First posted 2021-05-28 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Kidney Transplant; Complications; Diabetes Mellitus, Type 2
Keywords: Post operative kidney transplant
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Placebo-controlled, double-blind, randomized clinical trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I: With Type II Diabetes (Active Comparator): Kidney Transplant recipient with Type II diabetes, randomized to either Empagliflozin or a placebo.
  Interventions: Drug: Empagliflozin10Mg Tab; Drug: Placebo
- Arm 2: Without Diabetes (Active Comparator): Kidney Transplant recipient without Type II diabetes, randomized to either Empagliflozin or a placebo
  Interventions: Drug: Empagliflozin10Mg Tab; Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin10Mg Tab — Empagliflozin10 Mg daily or placebo daily for 18 months
Drug: Placebo — 10Mg Placebo Tab

SUMMARY:
CREST-KT is a single-center, double-blinded, randomized trial of empagliflozin therapy in 72 kidney transplant recipients with (n=36) and without type 2 diabetes (n=36). After evenly dividing patients by type 2 diabetes diagnosis, patients will be randomized 2:1 to empagliflozin 10mg versus placebo.

DETAILED DESCRIPTION:
A screening visit will occur at which time an informed consent will be obtained, and eligibility determined. Women of childbearing potential will have a serum pregnancy test performed. This will be followed by a baseline visit. A renal biopsy and a 3D echocardiogram will be performed. At the next visit randomization will be performed and the subjects will receive their study medication, either empagliflozin or a placebo. Following the randomization visit the subject will return every 3 months (visits 2-7) for a total of 6 visits spanning 18 months. At each visit vital signs and weight will be taken. Other procedures include labs drawn for hematology, basic chemistry, coagulation, Glycated hemoglobin and serum insulin. A 3 D echocardiogram is repeated on Visits 4 and 6. A renal biopsy is repeated on Visit 3.

ELIGIBILITY:
Inclusion Criteria:

1. Equal to or greater than 12 months and up tp 60 months post kidney transplant
2. Estimated glomerular filtration rate (eGFR) equal to or greater than 30ml/min/1.73m squared at screening
3. Standard immunosuppression, including calcineurin inhibitor, Mycophenolate Mofetil or Sodium and a glucocorticoid
4. Able to provide written consent -

Exclusion Criteria:

1. Type I diabetes
2. Any other solid organ transplant
3. Hemoglobin A1c greater than 12 %
4. SGLT2i use at the time of enrollment
5. Prior SGLT2i allergy or intolerance
6. Pregnant or nursing at the time of enrollment
7. History of antibody medicated rejection (AMR) or a Banff score greater than 2B for acute cellular rejection (ACR)
8. Active anticoagulant use other than aspirin 81 mg for primary prevention of cardiovascular disease
9. Known positive donor-specific antibodies prior to enrollment
10. Uncircumcised men
11. Greater than 2 urinary tract infections (UTI) over the 12 months prior to enrollment
12. Any genital infections over the 12 months prior to enrollment -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2026-01-22 (Actual); Study Completion 2026-01-22 (Actual)

PRIMARY OUTCOMES:
Change in kidney function as measured by eGFR | Baseline, 6 months, 9 months, 12 months and 18 months
  eGFR will be measured by blood test
Change in kidney function as measured by albuminuria | Baseline, 6 months, 9 months, 12 months and 18 months
  Albuminuria will be measured by urine Albumin/Creatinine Ratio
Change in cardiac structure | Baseline, month 9 and month15
  Cardiac structure as measured by the 3D echocardiogram
Change in blood insulin level | Baseline, month 6 and month 18
  Blood insulin level will be determined lab values
Change in fasting blood sugar | Baseline, month 6 and month 18
  Fasting Blood sugar will be determined lab values
Number of Urinary Tract infections | up to 18 months
  Data to be gathered from chart review and patient report
Number of Genital infections | up to 18 months
  Data to be gathered from chart review and patient report

SECONDARY OUTCOMES:
Change in kidney biopsy as measured by percentage of interstitial fibrosis | Baseline and 6 months
Changes in Hemoglobin A1C as measured by blood work | Baseline, Months 3,6,9,12,15 and 18

OTHER OUTCOMES:
Adverse events will be collected form the medical record and patient report | up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Myles Wolf, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared

REFERENCES:
- [Result] Stoumpos S, Jardine AG, Mark PB. Cardiovascular morbidity and mortality after kidney transplantation. Transpl Int. 2015 Jan;28(1):10-21. doi: 10.1111/tri.12413. Epub 2014 Aug 20. PMID 25081992
- [Result] Zinman B, Lachin JM, Inzucchi SE. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2016 Mar 17;374(11):1094. doi: 10.1056/NEJMc1600827. No abstract available. PMID 26981940
- [Result] Neal B, Perkovic V, Mahaffey KW, de Zeeuw D, Fulcher G, Erondu N, Shaw W, Law G, Desai M, Matthews DR; CANVAS Program Collaborative Group. Canagliflozin and Cardiovascular and Renal Events in Type 2 Diabetes. N Engl J Med. 2017 Aug 17;377(7):644-657. doi: 10.1056/NEJMoa1611925. Epub 2017 Jun 12. PMID 28605608
- [Result] Wiviott SD, Raz I, Bonaca MP, Mosenzon O, Kato ET, Cahn A, Silverman MG, Zelniker TA, Kuder JF, Murphy SA, Bhatt DL, Leiter LA, McGuire DK, Wilding JPH, Ruff CT, Gause-Nilsson IAM, Fredriksson M, Johansson PA, Langkilde AM, Sabatine MS; DECLARE-TIMI 58 Investigators. Dapagliflozin and Cardiovascular Outcomes in Type 2 Diabetes. N Engl J Med. 2019 Jan 24;380(4):347-357. doi: 10.1056/NEJMoa1812389. Epub 2018 Nov 10. PMID 30415602
- [Result] Halden TAS, Kvitne KE, Midtvedt K, Rajakumar L, Robertsen I, Brox J, Bollerslev J, Hartmann A, Asberg A, Jenssen T. Efficacy and Safety of Empagliflozin in Renal Transplant Recipients With Posttransplant Diabetes Mellitus. Diabetes Care. 2019 Jun;42(6):1067-1074. doi: 10.2337/dc19-0093. Epub 2019 Mar 12. PMID 30862658
- [Result] Heerspink HJ, Perkins BA, Fitchett DH, Husain M, Cherney DZ. Sodium Glucose Cotransporter 2 Inhibitors in the Treatment of Diabetes Mellitus: Cardiovascular and Kidney Effects, Potential Mechanisms, and Clinical Applications. Circulation. 2016 Sep 6;134(10):752-72. doi: 10.1161/CIRCULATIONAHA.116.021887. Epub 2016 Jul 28. PMID 27470878